CLINICAL TRIAL: NCT06100965
Title: The Effects of Reduced Dose Alemtuzumab for Severe Kidney Transplant Rejection
Brief Title: Reduced-dose Alemtuzumab for Kidney Transplant Rejection
Acronym: ROSETTE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lukas K. van Vugt, Research coordinator, Erasmus Medical Center
Other Study IDs: NL82152.078.23
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplant Rejection
Keywords: alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary samples Whole-blood and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, follow-up study of kidney transplant recipients treated with alemtuzumab anti-rejection therapy for severe or glucocorticoid-resistant kidney transplant rejection.

DETAILED DESCRIPTION:
Study design: Prospective observational cohort study. Study population: Adult patients who are treated with alemtuzumab for severe or glucocorticoid-resistant kidney transplant rejection.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: Lymphocyte (subtype) repopulation, serious infections, one-year graft survival, alemtuzumab plasma levels, intra-cellular signalling of repopulated T and B cells, cytokine-levels, donor-specificity of repopulated T cells, differences pre- and post-treatment of donor-derived cell-free DNA, plasma nucleosomes, urinary chemokines, urinary extracellular vesicles, breath-pattern analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Treatment for severe or glucocorticoid-resistant kidney transplant rejection with alemtuzumab.

Exclusion Criteria:

* Treatment with a different lymphocyte depleting agent (e.g. rATG) prior to treatment with alemtuzumab for the same rejection episode.
* Recipients who have T cell counts below 200 × 106/L before the start of therapy (for instance, because of lymphocyte depleting induction therapies).
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients who experience severe or glucocorticoid-resistant rejection of their allograft.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with lymphocyte repopulation | 6 months and 1 year
  Outcome reporting of the proportion of patients that has repopulation of T and B lymphocytes, defined as cell counts of >200 10E6/L for T lymphocytes and > 100 10E6/L for B lymphocytes.

SECONDARY OUTCOMES:
Cumulative incidence of graft loss | 6 months, 1 year
  Cumulative incidence of graft loss at specified time-points with death as competing risk, computed by cumulative incidence functions.
Serious infections | 6 months, 1 year
  Necessitating hospital admission, or hospital-acquired
Patient survival | 6 months, 1 year
  Proportion of patients who survived at specified time-points, computed with kaplan-meier estimates at specified time-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided